CLINICAL TRIAL: NCT02237417
Title: A Randomized, Open Label, Parallel Group, Study of the Impact of Aripiprazole (Abilify®) Once Monthly Versus Standard of Care Oral Antipsychotic Medications on Changes in Brain Structure and Metabolism
Brief Title: Impact of Aripiprazole Once Monthly Medications on Changes in Brain Structure and Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00073657
Record Dates: First submitted 2014-09-03; First posted 2014-09-11 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
Keywords: MRI; Imaging; Antipsychotic
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Control (Other): Healthy individuals with no mental health diagnosis
  Interventions: Other: No Treatment
- Individuals with Schizophrenia (Group A) (Active Comparator): Individuals with a diagnosis of Schizophrenia undergoing standard of care treatments.
  Interventions: Drug: Standard of Care Oral antipsychotics
- Individuals with Schizophrenia (Group B) (Active Comparator): Individuals with Schizophrenia who are receiving treatment with Aripiprazole once monthly injections.
  Interventions: Drug: IM aripiprazole once monthly

INTERVENTIONS:
Drug: Standard of Care Oral antipsychotics — A total of 15 to 20 subjects with schizophrenia will receive SOC oral antipsychotic medications (e.g., aripiprazole (Abilify®), risperidone (Risperdal®), lurasidone HCI (Latuda®), quetiapine fumarate (Seroquel®), olanzapine (Zyprexa®), and ziprasidone HCI(Geodon®)) or once monthly aripiprazole (Abilify®), PO daily, in accordance with their respective product labeling.
  Arms: Individuals with Schizophrenia (Group A)
Drug: IM aripiprazole once monthly — A total of 30 to 40 subjects with schizophrenia will receive aripiprazole (Abilify®) monthly, at a starting dose of 400 mg IM or an approved dose based on the investigator's judgment and in accordance with product labeling.
  Arms: Individuals with Schizophrenia (Group B)
Other: No Treatment — A total of 15 healthy controls will participate in the study and will not receive medication
  Arms: Healthy Control

SUMMARY:
This is a Phase 4, randomized, open-label, parallel group study designed to assess the clinical and biological effects of 12 months of treatment with long acting intramuscular (IM) aripiprazole (Abilify®) as measured by clinical and behavioral measures, and changes on magnetic resonance imaging (MRI) scans in subjects with schizophrenia compared with SOC oral antipsychotic medications and compared with a healthy control group.

DETAILED DESCRIPTION:
This is a Phase 4, randomized, open-label, parallel group study designed to assess the clinical and biological effects of 12 months of treatment with long acting intramuscular (IM) aripiprazole (Abilify®) as measured by clinical and behavioral measures, and changes on magnetic resonance imaging (MRI) scans in subjects with schizophrenia compared with SOC oral antipsychotic medications and compared with a healthy control group.

It is hypothesized that improved treatment compliance will lead to fewer white matter changes in the brain. Fewer white matter changes will be demonstrated via neuroimaging as increased FA and BPF values in the prefrontal region, and an increase in metabolites in a voxel centered on the anterior cingulate cortex (ACC) as seen with MRS. Therefore, the aim of this study is to examine the structural and metabolic effects of aripiprazole (Abilify®) once monthly in patients with schizophrenia using MRI techniques and to examine these effects in association with cognitive and clinical measures.

ELIGIBILITY:
Inclusion Criteria for All Subjects

* Are able to provide written informed consent.
* Are male and female subjects 18 to 35 years of age, inclusive, at time of informed consent.

Inclusion Criteria for Subjects with Schizophrenia

* Have a current diagnosis of schizophrenia as defined by DSM IV-TR criteria and a history of the illness for at least 1 year prior to screening and at least two prior psychotic episodes based on medical records or a qualified and reliable health care provider.
* Require, in the investigator's judgment, chronic treatment with an antipsychotic medication.
* Are able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, IM depot injection, and discontinuation of prohibited concomitant medications, read and understand the written word in order to complete subject-reported outcomes measures, and be reliably rated on assessment scales.
* Are male and female subjects who are surgically sterile (i.e., have undergone orchiectomy or hysterectomy, respectively; female subjects who have been postmenopausal for at least 12 consecutive months; or male and female subjects who agree to remain abstinent or to practice double barrier forms of birth control from trial screening through 30 days (for females) and 90 days (for males) from the last dose of IMP for SOC oral antipsychotics and 150 days for females and 180 days for males for aripiprazole depot. If employing birth control, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pill, birth control implant, birth control depot injections, condom, or sponge with spermicide.

Exclusion Criteria All Subjects

* Presence of any metal implants, pacemakers, unremovable prosthetic device, or other device or situation that may preclude imaging
* History of a head injury with loss of consciousness > 5 minutes
* Has a significant medical condition that would expose the subject to undue risk or interfere with study assessments.

Exclusion Criteria for Subjects with Schizophrenia

* Has a current DSM-IV-TR diagnosis other than schizophrenia, including schizophreniform disorder, schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also excluded are subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Is considered resistant/refractory to antipsychotic treatment by history (failed two prior antipsychotic medication trials) or response only to clozapine.
* Has a significant risk of violent behavior or a significant risk of committing suicide based on history or investigator's discretion.
* Has met DSM-IV-TR criteria for any significant substance use disorder within 3 months prior to screening, excluding caffeine, nicotine, or marijuana.
* Is known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones, or hypersensitivity to antipsychotic agents, including aripiprazole.
* Has a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia at screening per the investigator's discretion.
* Has a history of seizures or any other medical condition that would expose the subject to undue risk or interfere with study assessments.
* Is involuntarily incarcerated.
* Has undergone electroconvulsive therapy in the 2 years prior to enrollment in the study.
* Has used an investigational agent or has participated in a clinical study with aripiprazole IM depot or any other antipsychotic depot preparation within 30 days of screening.
* Has clinically significant abnormalities in laboratory test results, vital signs, or ECG results.
* Requires more than one benzodiazepine beyond screening (e.g., lorazepam and oxazepam).
* Fails to washout from prohibited concomitant medications, including the use of or CYP3A4 inducers, a second antipsychotic, antidepressants (including monoamine oxidase inhibitors), and mood stabilizers.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Yurgelun-Todd, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Control | Individuals With Schizophrenia (Group A) | Individuals With Schizophrenia (Group B)
Started | 16 | 15 | 16
Completed | 16 | 9 | 7
Not Completed | 0 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Individuals With Schizophrenia (Group A) | Individuals With Schizophrenia (Group B) | Total
Number analyzed (Participants) | 16 | 15 | 16 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 16 | 47
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 28 [18 to 50] | 30 [18 to 50] | 28 [18 to 50] | 28 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 3 | 14
  Male | 10 | 10 | 13 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 5 | 14
  Not Hispanic or Latino | 14 | 8 | 10 | 32
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in Fractional Anisotropy (FA)
Description: To determine if there are differences in prefrontal white matter fractional anisotropy (FA) in subjects with schizophrenia from baseline at 12 months of treatment with aripiprazole (Abilify®) once monthly compared with standard of care (SOC) oral antipsychotic medications (e.g., aripiprazole (Abilify®), risperidone (Risperdal®), lurasidone HCI (Latuda®), quetiapine fumarate (Seroquel®), olanzapine (Zyprexa®), and ziprasidone HCI (Geodon®)).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Control | Individuals With Schizophrenia (Group A) | Individuals With Schizophrenia (Group B)
Number analyzed (Participants) | 16 | 15 | 16
Participants | 13 | 9 | 7

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Three types of adverse event data are to be reported: "All-Cause Mortality," "Serious," and "Other (Not Including Serious)" Adverse Events.
Arm/Group | Healthy Control | Individuals With Schizophrenia (Group A) | Individuals With Schizophrenia (Group B)
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/9 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/16 | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-07-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT02237417/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT02237417/ICF_001.pdf